CLINICAL TRIAL: NCT07015866
Title: Effects of Creative Arts Therapy on Body Image, Self-esteem, Anxiety and Depression in Men With Prostate Cancer After Active Treatment: A Feasibility Randomised Controlled Trial
Brief Title: Creative Arts Therapy on Body Image, Self-esteem, Anxiety and Depression in Post-Treatment Prostate Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); University of Derby (Other)
Responsible Party: Principal Investigator, ABU ODAH, Hammoda MM, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22231641
Record Dates: First submitted 2025-05-23; First posted 2025-06-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Creative Arts Therapy
Keywords: creative arts therapy; prostate cancer; body image; slef-esteem; anxiety; depression; active treatment
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative arts therapy (Experimental): The intervention will be offered throughout five sessions. Session themes are as follows: 'bridge drawing', 'analogue drawing', 'life-sized body outline', a 'free session' to allow patients to express their feelings, and a final review with the art therapist in which all sessions will be brought to a conclusion. The first individual session, 'bridge drawing', will be used to introduce the creative arts therapy approach and to elaborate on this project. The four other sessions will be group-based (with four participants per group), providing a supportive and communal environment where participants can engage in creative expression alongside others who may have had similar experiences or challenges. A session will be conducted each week over five weeks, with each session lasting 60 minutes. All sessions will be conducted in a room in the Urology Centre that has been equipped and prepared for the intervention.
  Interventions: Other: Creative arts therapy
- Guided group discussions (Active Comparator): Participants will engage in guided group discussions over five sessions. Each session will include a guided discussion focusing on self-care topics such as sleep hygiene, dental hygiene, nutrition, and personal interests and hobbies. The first individual session, 'Sleep hygiene, will be used to educate the participants of the importance of sleep and strategies to improve sleep quality. The four other sessions will be group-based (with four participants per group), focusing on dental hygiene, nutrition, personal interests and hobbies and general well-being and reflection. A session will be conducted each week over five weeks, with each session lasting 60 minutes. All sessions will be conducted in a room in the Urology Centre.
  Interventions: Other: Guided therapy group

INTERVENTIONS:
Other: Guided therapy group — Participants will engage in guided group discussions over five sessions. Each session will include a guided discussion focusing on self-care topics such as sleep hygiene, dental hygiene, nutrition, and personal interests and hobbies. The first individual session, 'Sleep hygiene, will be used to educate the participants of the importance of sleep and strategies to improve sleep quality. The four other sessions will be group-based (with four participants per group), focusing on dental hygiene, nutrition, personal interests and hobbies and general well-being and reflection. A session will be conducted each week over five weeks, with each session lasting 60 minutes. All sessions will be conducted in a room in the Urology Centre.
  Arms: Guided group discussions
Other: Creative arts therapy — The intervention will be offered throughout five sessions. Session themes are as follows: 'bridge drawing', 'analogue drawing', 'life-sized body outline', a 'free session' to allow patients to express their feelings, and a final review with the art therapist in which all sessions will be brought to a conclusion.
  The first individual session, 'bridge drawing', will be used to introduce the creative arts therapy approach and to elaborate on this project. The four other sessions will be group-based (with four participants per group), providing a supportive and communal environment where participants can engage in creative expression alongside others who may have had similar experiences or challenges. A session will be conducted each week over five weeks, with each session lasting 60 minutes. All sessions will be conducted in a room in the Urology Centre that has been equipped and prepared for the intervention.
  Arms: Creative arts therapy

SUMMARY:
The goal of this clinical study is to assess the feasibility of implementing a creative arts therapy intervention of drawing and painting in Hong Kong prostate cancer patients and preliminarily examine the effects of this intervention on prostate cancer patients' health outcomes via a two-armed randomized controlled trial. The two arms will be (i) the creative arts therapy intervention group and (ii) a active control group.

Participants will join five sessions. Sessions will start with a 10-15-minute rapport-building discussion and continue with a 60-minute intervention. Session themes are as follows: 'bridge drawing', 'analogue drawing', 'life-sized body outline', a 'free session' to allow patients to express their feelings, and a final review with the art therapist in which all sessions will be brought to a conclusion. Each session will follow a three-step process of psychodynamic model to ensure the optimal effect of the intervention. The interventions will be held at private room at hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants diagnosed with localised prostate cancer, regardless of the stage and age 18 years or older;
* are not currently receiving active therapy, including chemotherapy, radiotherapy or surgical treatment, by the time of the study or completed treatment more than one year ago and are not on any active treatment;
* were being followed up by the urology team or Department of Surgery at the Chinese University of Hong Kong;
* are willing to participate in the study;
* are able to read Chinese and communicate in Cantonese;
* are physically able to attend and complete art therapy sessions;
* do not have significant comorbidities, including cerebrovascular accident, severe depression, or dementia that could affect their ability to participate in the study;
* signed an informed consent form.

Exclusion Criteria:

* Adult participants diagnosed with a mixed type of terminal cancer;
* are undergoing active therapy;
* have participated in other art therapy interventions;
* have physical issues preventing them from holding a pen;
* have a mental status and/or communication problem that might compromise their capacity to give informed consent;
* have significant comorbidities such as cerebrovascular accident, severe depression, or dementia, as determined by standardized screening tools a score of 20-27 on the Patient Health Questionnaire and score 25 or less on the Mini-Mental State Examination.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Body image | Baseline and 5 weeks
  The Chinese version of the 10-item Body Image Scale (BIS) will be used to assess participants' perception of their body image, including influence, actions and cognition. Each item is scored on a 4-point scale ranging from 0 (not at all) to 3 (very much). The BIS overall summary score ranges from 0 to 30, with a higher score indicating a poorer body image. The BIS was translated by school of nursing team at the Hong Kong Polytechnic University and has been utilised by our team
Self-esteem | Baseline and 5 weeks
  The Chinese version of the Rosenberg Self-Esteem Scale (RSES) will be used to evaluate participants' general self-esteem. It consists of 10 items assessing positive and negative feelings about the self. Each item is scored on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The RSES overall score ranges from 10 to 40, with a higher score indicating high self-esteem. The RSES version as translated by school of nursing team at the Hong Kong Polytechnic University and has been utilised by our team.
Anxiety and depression | Baseline and 5 weeks
  The Chinese version of the Hospital Anxiety and Depression Scale (HADS) will be used to assess participants' anxiety and depression levels. The HADS consists of 14 items categorised into two subscales: anxiety and depression. Scores for each subscale are calculated and classified into one of three categories: normal cases (scores of 0-7), borderline cases (scores of 8-10) and cases (scores of 11-21). The Chinese version of the HADS has a strong intercorrelation between anxiety and depression in cancer patients (r = 0.83).
Retention rate | Baseline, 5 weeks and 3 months post
  The number of patients who remain in the study divided by the number of patients randomised. The retention rate will be calculated for each arm at baseline and follow-ups.